CLINICAL TRIAL: NCT07209540
Title: European LUpuS Inception-Cohort Developing initiATivE
Acronym: ELUSIDATE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 36-18-2025
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: lupus; systemic lupus erythematosus; SLE; treat-to-target; prediction
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — EDTA plasma, Serum, PBMCs, PAX gene tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn more about how systemic lupus erythematosus (SLE or lupus) develops in the first years after diagnosis, and how patients respond to different treatments.

The main questions the study aims to answer are:

How many patients with newly diagnosed lupus reach remission or low disease activity in the first years after starting treatment?

Which biological markers (in blood or urine) can help predict treatment response, disease complications, or symptoms such as pain and fatigue?

Adults recently diagnosed with lupus (within the past 6 months) will be invited to participate. They will continue with their normal medical care, but in addition, they will take part in study visits over a 5-year period. At these visits, doctors will collect information about symptoms, treatment, and quality of life. Blood and urine samples will also be stored in a biobank for later analysis.

Around 720 patients from several European countries are expected to join the study. Because participants are included very soon after diagnosis, researchers can follow the course of lupus from the beginning, before long-term treatment or damage occurs.

By combining clinical information and biological samples, researchers hope to identify new ways to understand lupus, improve treatment strategies, and eventually develop personalized medicine approaches. This could help future patients achieve better disease control, fewer complications, and improved quality of life.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

1. Introduction Systemic lupus erythematosus (SLE) is a complex autoimmune disease with diverse clinical manifestations. Despite recent therapeutic advances, challenges persist, including increased mortality, long-term complications, and impaired quality of life. We still use a step-up approach to treatment guided by EULAR recommendations although we know only around 50% of patients reach a low disease activity state within a year.

   The establishment of a European inception cohort with a biobank aims to address these challenges by providing standardized data, particularly in the context of evolving treatment paradigms.
2. Background and Rationale SLE's heterogeneity poses challenges, and global cohorts face variability in patient management and genetic diversity. A European inception cohort offers advantages, including homogeneity in treatment standards and genetic backgrounds, enhancing data reliability. Recent therapeutic approvals signal progress, with a shift towards a "treat-to-target" approach, underscoring the need for a more nuanced understanding of disease activity and response factors.
3. Objectives The primary objective is to establish a European, multi-national, prospective, observational inception SLE cohort with a comprehensive biobank.

   The study aims to assess the frequency of SLE patients achieving remission or low disease activity using novel criteria within specific timeframes.

   Utilizing the biobank, the study aims to identify novel biomarkers associated with treatment response/non-response, SLE-related comorbidities, pain, fatigue, and genetic factors. These objectives include investigating soluble biomarkers, genetic associations, metabolites, and risk factor algorithms that contribute to understanding disease mechanisms, treatment responses, and the development of comorbidities.
4. Study Design This European, multi-national, multi-centric, prospective, observational inception cohort involves follow-up visits at baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years. The study design encompasses a main protocol, a biobanking module, and optional subprotocols to address specific research questions.
5. Methods Adult patients with clinical diagnosis of SLE and fulfilling the 2019 ACR/EULAR criteria before initiation treatment are eligible. If treatment has been initiated, patients can still be included if it is less than six months since diagnosis and the patient has clinically and biochemically active disease (SLEDAI>6). Recruitment will take place over a two-year enrolment period and a five-year follow-up period, with an estimated 720 patients enrolled. Blood samples will be stored locally and later transferred to a centralized coordinating center. Clinical data, PROMs, blood, and urine will be collected at each visit.
6. Perspective This protocol aims to propel SLE research forward, providing a robust foundation for understanding the disease, its treatment, and factors influencing patient outcomes. Through a collaborative, multi-national effort, this initiative endeavors to pave the way for personalized medicine in the management of systemic lupus erythematosus.
7. Novelty To date, the SLICC SLE baseline cohort is the only existing international baseline cohort. It was initiated in 1998 and has generated significant new knowledge in the field of lupus over the past 25 years. The SLICC inception cohort was developed to better understand atherosclerosis, nervous system involvement, lupus nephritis and damage accumulation and their economic impact. It includes patients within 15 months of diagnosis and recruitment was completed in 2011. Since then, much progress has been made in the management of SLE. The re-enlistment of an inception cohort can help to assess the practical implementation and impact of new trends in diagnosis and treatment, as well as their effect on disease progression and outcome. ELUSIDATES aims to enroll patients immediately after diagnosis to ensure a true inception cohort. Ideally, patients will have no prior treatment or damage and can be followed for the first 5 years of the disease. In addition to clinical data, and in contrast to the SLICC inception cohort, biosampling will allow characterization of patients at the molecular level and analysis of biomarkers and predictive models.

Recruitment will be incentivised by allowing participating centres to submit their research sub-protocols, a strategy to ensure high recruitment rates.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion at clinical diagnosis of SLE (or strong clinical suspicion hereof) before initiating treatment (if treatment has been initiated, patients can still be included if it is less than six months since diagnosis and the patient has clinically and biochemically active disease (SLEDAI>6).
* Fulfilling the 2019 ACR/EULAR criteria for Systemic Lupus Erythematosus
* >18 years of age (adult onset SLE)
* Ability to provide informed voluntary consent.

Exclusion Criteria:

* Diagnosed with overlapping systemic autoimmune diseases other than secondary Sjögren's syndrome or antiphospholipid syndrome.
* Active treatment for malignancy at the time of enrolment, except for non-melanoma skin cancer or localized carcinoma in situ of the skin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with a new diagnosis of systemic lupus erythematosus (SLE) according to the 2019 ACR/EULAR criteria. Patients must be treatment-naïve. If they have started treatment they must have clinically and biochemically active disease. Approximately 700 participants will be enrolled across multiple European centers.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2033-07-01 (Estimated)

PRIMARY OUTCOMES:
DORIS remission | 1 year
  How many patients achieve DORIS remission 1 year after diagnosis
Lupus Low Disease Activity | 1 year
  How many patients have achieved LLDAS at 1 year after diagnosis

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected during the trial will be shared with qualified researchers after completion of the study and publication of the primary results. Data access will be provided upon submission of a methodologically sound proposal, subject to approval by the study steering committee and compliance with ethical and legal regulations.
Supporting Information: Study Protocol
Time Frame: Protocol and data will be available from completion of inclusion and minimum 5 years after study end.
Access Criteria: Access will be granted for scientifically sound proposals addressing questions related to lupus, treatment outcomes, or biomarkers. Requests must be submitted to the study steering committee for review and approval. Approved researchers will sign a data access agreement and receive data through a secure, controlled-access platform.